CLINICAL TRIAL: NCT04841473
Title: Popular Opinion Leaders as a Sports Concussion Prevention Strategy in Middle Schools-The TRAIN Study, a Randomized Control Study
Brief Title: The TRAIN Study: A Concussion Prevention Strategy in Middle Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-0314
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: Concussion, Brain
Keywords: Concussion; Prevention; Management
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Concussion Education (Active Comparator): Participants will receive standard concussion education materials (online training) focused on concussion prevention in youth sport.
  Interventions: Other: Standard Concussion Education
- TRAIN Concussion Education (Experimental): After receiving the standard concussion education materials (online training), participants will receive an additional module, the TRAIN concussion education module.
  Interventions: Other: TRAIN Concussion Education

INTERVENTIONS:
Other: TRAIN Concussion Education — Participants will receive the TRAIN concussion education module.
  Arms: TRAIN Concussion Education
Other: Standard Concussion Education — Participants will receive a standard concussion education module.
  Arms: Standard Concussion Education

SUMMARY:
Purpose: The purpose of this study is to evaluate the effectiveness of a theory-driven intervention (TRAIN concussion education) to improve parental concussion-related attitudes, beliefs, intentions, confidence in knowledge, and self-efficacy.

Participants: 180 parents of United States middle school aged children whose children have been engaged in organized sports within the past 2 years.

Procedures: The study is a single-blind (participants) randomized control trial. The investigators will randomize eligible parents into two groups: (1) control (standard concussion education); and treatment (standard concussion education AND TRAIN concussion education) to evaluate the effectiveness of the TRAIN concussion education intervention.

DETAILED DESCRIPTION:
A convenience sample of participants will be recruited from parents of United States middle school aged children whose children have been engaged in organized sports within the past 2 years. Interested parents will contact study stuff, who will ensure eligibility criteria are met.

Upon this, and completing the written informed consent process, participants will be assigned a unique identifier and randomized (simple) without replacement to one of the two study arms (control vs. treatment), using a predetermined random number generator in Excel.

Participants in the control group will receive standard concussion education materials focused on concussion prevention in youth sport. Participants in the treatment group will receive the same standard concussion education materials AND the TRAIN concussion education module. The TRAIN education module is grounded in a theoretical structure inclusive of the original intervention tenants of the Popular Opinion Leader (POL) and Diffusion of Innovations frameworks, and within the context of the socioecological model.

Participants will complete a self-administered online pre-test survey, which includes assessments of concussion-related attitudes, beliefs, intentions, confidence in knowledge, and self-efficacy. After completion of the pre-test survey, participants will complete their assigned intervention (TRAIN concussion education module + standard concussion education materials versus standard concussion education materials only).

Upon completion of their assigned intervention, participants will complete the online survey again to obtain post-test measures (post-test survey). Participants will also be scheduled to complete individual semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* Adult with a child/children enrolled in a United States middle school
* Adult whose child has participated in organized sports in the past 2 years

Exclusion Criteria:

• Adult without a child/children enrolled in a United States middle school

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Concussion-Related Beliefs Change Score | Baseline (pre-intervention) and follow-up (post intervention approximately 7-30 days after intervention completion)
  Participants are asked 6 questions concerning beliefs related to concussion risk, symptoms, and management. These items are added together to compute an overall score. Scoring scale ranges from a minimum of 6 to a maximum 24, where a higher score indicated more favorable beliefs. A change score will be computed post score-pre score.
Concussion-Related Attitudes Change Score | Baseline (pre-intervention) and follow-up (post intervention approximately 7-30 days after intervention completion)
  Participants are asked 20 survey items identifying an individual's attitudes about a certain behavior (e.g., seeking care). Each item is added together to compute an overall attitude score. Scoring scale ranges from a minimum of 20 to a maximum of 140, where higher scores indicate more favorable attitudes. A change score will be computed post score-pre score.

SECONDARY OUTCOMES:
Confidence in Concussion-Related Knowledge Change Score | Baseline (pre-intervention) and follow-up (post intervention approximately 7-30 days after intervention completion)
  Participants are asked 2 questions concerning confidence in knowing and recognizing concussion symptoms. These items are added together to compute an overall score. Scoring scale ranges from a minimum of 2 to a maximum 8, where a higher score indicated better confidence in concussion knowledge. A change score will be computed post score-pre score.
Concussion-Related Intentions Change Score | Baseline (pre-intervention) and follow-up (post intervention approximately 7-30 days after intervention completion)
  Participants are asked 4 questions assessing intention to engage in or talk with others about concussion prevention. The items are totaled to compute an overall behavioral intention score. Scoring scale ranges from a minimum of 4 to a maximum of 16, where a higher score indicates a better likelihood to engage in favorable behaviors related to concussion prevention. A change score will be computed post score-pre score.
Concussion-Related Self-Efficacy Change Score | Baseline (pre-intervention) and follow-up (post intervention approximately 7-30 days after intervention completion)
  Participants are asked 8 questions assessing their self-efficacy regarding engaging in or talking with others about concussion prevention. The items are totaled to compute an overall self-efficacy score. Scoring scale ranges from a minimum of 8 to a maximum of 32, where a higher score indicates higher self-efficacy. A change score will be computed post score-pre score.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Kerr, PhD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Injury Prevention Research Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP
Time Frame: 9 - 36 months following publication
Access Criteria: IRB, IEC, or REB and an executed data use/sharing agreement with the University of North Carolina at Chapel Hill

DOCUMENTS (1):
  • Informed Consent Form (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/73/NCT04841473/ICF_000.pdf